CLINICAL TRIAL: NCT06250387
Title: Prospective Feasibility Study of Endobronchial Ultrasound Transbronchial Cryobiopsy (EBUS-TBCB 1.1 mm Probe) Among Patients With Mediastinal Lymphadenopathies
Acronym: EBUS-CRYO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A00969-36
Record Dates: First submitted 2024-01-12; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Endobronchial Mass
Keywords: Patients with mediastinal lymphadenopathies.

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with mediastinal lymphadenopathy (Experimental): Patients with suspicion of lymphoma, sarcoidosis and tuberculosis, presenting with mediastinal lymphadenopathy confirmed by a CT scan and/ or PET scan and patients with previous negative EBUS-TBNA.
  Interventions: Procedure: Endobronchial ultrasound transbronchial cryobiopsy

INTERVENTIONS:
Procedure: Endobronchial ultrasound transbronchial cryobiopsy — Endobronchial Ultrasound (EBUS) :
  EBUS is usually performed under general anesthesia using a laryngeal masque. It has a linear ultrasonography with a 7.5 MHz frequency. The distal part of the endoscope contains a water filled balloon used as a liquid interface, camera, light source and a working channel. The needle is protected by a sheath to prevent working channel damage. The endoscope is connected to a processor that reflects both endobronchial and ultrasound images on a screen.
  EBUS - TBNA : EBUS - Transbronchial needle aspiration EBUS - TBCB: EBUS - Transbronchial Cryo Biopsy
  Other Names: Endobronchial ultrasound transbronchial cryobiopsy (EBUS-TBCB 1.1 mm probe) among patients with mediastinal lymphadenopathies.

SUMMARY:
Mediastinal lymph nodes enlargement with short axis diameter >15 mm is conventionally defined as a mediastinal lymphadenopathy. The causes of mediastinal lymphadenopathy can be malignant or benign, (infectious, inflammatory, and other such as drug toxicity).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age
* Mediastinal and/or hilar lymphadenopathies > 20 mm on an injected chest CT scan
* Suspicion of lymphoproliferative disease, sarcoidosis or tuberculosis
* Hypermetabolism of mediastinal and/or hilar lymphadenopathies on PET scan (SUV max > 3)
* No contraindication for general anesthesia
* French-speaking Patient
* -Signed informed consent

Exclusion Criteria:

* Patient not covered by the French social security system
* Patient with legal protection
* Pregnant or breastfeeding patient (if applicable)
* Patient under guardianship or curatorship
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of EBUS TBCB 1.1 mm probe. | 6 Months
  Number of successes of the procedure. A success is defined by the ability to perform a biopsy.

SECONDARY OUTCOMES:
To estimate the sensitivity of EBUS TBCB probe 1.1 mm in the diagnosis of mediastinal lymphadenopathy. | 7 Months
  anapathology analysis
To estimate the specificity of EBUS TBCB probe 1.1 mm in the diagnosis of mediastinal lymphadenopathy. | 7 Months
To estimate the procedure time. | Day 0
  The procedure time is defined by the time elapsed between introduction and removal of the EBUS probe
To assess the post-procedure complications rate. | 1 Month

REFERENCES:
- [Background] Ernst A, Anantham D, Eberhardt R, Krasnik M, Herth FJ. Diagnosis of mediastinal adenopathy-real-time endobronchial ultrasound guided needle aspiration versus mediastinoscopy. J Thorac Oncol. 2008 Jun;3(6):577-82. doi: 10.1097/JTO.0b013e3181753b5e. PMID 18520794
- [Background] Silvestri GA, Gonzalez AV, Jantz MA, Margolis ML, Gould MK, Tanoue LT, Harris LJ, Detterbeck FC. Methods for staging non-small cell lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e211S-e250S. doi: 10.1378/chest.12-2355. PMID 23649440